CLINICAL TRIAL: NCT04316754
Title: Effectiveness of Music During Cardiac Catheterization On Children's Pain, Fear, Anxiety and Vital Signs: A Randomized, Double-Blind Controlled Trial
Brief Title: Effectiveness of Music During Cardiac Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Research Assistant, Faculty of Health Sciences, Department of Pediatric Nursing, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019/369
Record Dates: First submitted 2020-03-09; First posted 2020-03-20 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Angiography
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No music will be played to the control group.
- Intervention 1 (Active Comparator): During angiography, the Intervention-1 group will listen to the music that the child wants to listen.
  Interventions: Other: music
- Intervention-2 (Active Comparator): The Intervention-2 group will listen to the music which determined by the researchers. The music which determined by the researchers is "The art of fugue" by Johann Sebastian Bach. The music to be played has been decided by examining the literature. (DOI: 10.4274/jpr.24892)
  Interventions: Other: music

INTERVENTIONS:
Other: music — During angiography, the Intervention-1 group will listen to the music that the child wants to listen to. The Intervention-2 group will listen to the "Arts of Fugue" by Bach. No music will be played to the control group.
  Arms: Intervention 1; Intervention-2

SUMMARY:
The research was planned on a randomized controlled experimental basis. Simple stratified randomization will be performed according to gender and age. Consent will be obtained from children and parents who agree to participate in the research.

Before angiography, "Child Fear Scale", "State-Trait Anxiety Scale (STAI-TX)", and "Vital Signs Follow-up Form" will be applied to all children taking part in the study and life signs will be recorded.

During angiography, the first group will listen to the music that the child wants to listen to. The second group will listen to the music which determined by the researchers. No music will be played to the control group. During angiography (when the child is listening to the music) vital signs will be recorded in 0. min., 1st minute, 5th minute, 10th minute, 15th minute, 30th minute and 60th minute.

"Numerical Pain Scale", "Child Fear Scale", "State Anxiety Scale", and "Vital Signs Follow-up Form" will be re-evaluated to all three groups after angiography.

DETAILED DESCRIPTION:
This study was planned to determine the effect of music during angiography on pain, fear, anxiety and life signs in children aged 7-18.

The research was planned on a randomized controlled experimental basis. Simple stratified randomization will be performed according to gender and age. Consent will be obtained from children and parents who agree to participate in the research.

Before angiography, "Child Fear Scale", "State-Trait Anxiety Scale (STAI-TX)", and "Vital Signs Follow-up Form" will be applied to all children taking part in the study and life signs will be recorded.

The sample size of the study was determined and the effect size was 0.25 based on the Standard effect sizes determined by Cohen. In the study, the sample number of 0.84 in the statistical power α=0.05 confidence interval was calculated as 36 for each group.

During angiography, the first group will listen to the music that the child wants to listen to. The second group will listen to the music which determined by the researchers. No music will be played to the control group. During angiography (when the child is listening to the music) vital signs will be recorded in 0. min., 1st minute, 5th minute, 10th minute, 15th minute, 30th minute and 60th minute.

"Numerical Pain Scale", "Child Fear Scale", "State Anxiety Scale", and "Vital Signs Follow-up Form" will be re-evaluated to all three groups after angiography.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Being between 7-18 years of age
* Lack of communication problems (vision, hearing, mental)
* Being informed about surgical intervention
* Lack of prior surgical intervention experience
* Receiving sedoanalgesia during angiography

Exclusion Criteria:

* Intubation of the child during angiography
* Parent's refusal to take part in the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
child's heart rate | baseline (at the beginning of angiography)
  the child's pulse rate will be measured.
child's heart rate | 1st minute of the angiography
  the child's pulse rate will be measured.
child's heart rate | 5th minute of the angiography
  the child's pulse rate will be measured.
child's heart rate | 10th minute of the angiography
  the child's pulse rate will be measured.
child's heart rate | 30th minute of the angiography
  the child's pulse rate will be measured.
child's heart rate | 60th minute of the angiography
  the child's pulse rate will be measured.
child's respiratory rate | Baseline (at the beginning of angiography)
  the child's respiratory rate will be measured.
child's respiratory rate | 1st minute of the angiography
  the child's respiratory rate will be measured.
child's respiratory rate | 5th minute of the angiography
  the child's respiratory rate will be measured.
child's respiratory rate | 10th minute of the angiography
  the child's respiratory rate will be measured.
child's respiratory rate | 15th minute of the angiography
  the child's respiratory rate will be measured.
child's respiratory rate | 30th minute of the angiography
  the child's respiratory rate will be measured.
child's respiratory rate | 60th minute of the angiography
  the child's respiratory rate will be measured.
child's blood pressure | baseline (at the beginning of angiography)
  the child's blood pressure will be measured.
child's blood pressure | 1st minute of the angiography
  the child's blood pressure will be measured.
child's blood pressure | 5th minute of the angiography
  the child's blood pressure will be measured.
child's blood pressure | 10th minute of the angiography
  the child's blood pressure will be measured.
child's blood pressure | 15th minute of the angiography
  the child's blood pressure will be measured.
child's blood pressure | 30th minute of the angiography
  the child's blood pressure will be measured.
child's blood pressure | 60th minute of the angiography
  the child's blood pressure will be measured.
child's body temperature | Baseline (at the beginning of angiography)
  the child's body temperature will be measured.
child's body temperature | 1st minute of the angiography
  the child's body temperature will be measured.
child's body temperature | 5th minute of the angiography
  the child's body temperature will be measured.
child's body temperature | 10th minute of the angiography
  the child's body temperature will be measured.
child's body temperature | 15th minute of the angiography
  the child's body temperature will be measured.
child's body temperature | 30th minute of the angiography
  the child's body temperature will be measured.
child's body temperature | 60th minute of the angiography
  the child's body temperature will be measured.
child's oxygen saturation | baseline (at the beginning of angiography)
  the child's oxygen saturation will be measured.
child's oxygen saturation | 1st minute of the angiography
  the child's oxygen saturation will be measured.
child's oxygen saturation | 5th minute of the angiography
  the child's oxygen saturation will be measured.
child's oxygen saturation | 10th minute of the angiography
  the child's oxygen saturation will be measured.
child's oxygen saturation | 15th minute of the angiography
  the child's oxygen saturation will be measured.
child's oxygen saturation | 30th minute of the angiography
  the child's oxygen saturation will be measured.
child's oxygen saturation | 60th minute of the angiography
  the child's oxygen saturation will be measured.
child's fear | up to 60 min (when the child wakes up from anaesthetic)
  Child fear will be assessed by "Children's Fear Scale". This scale includes 5 different facial expressions. This scale is rated from 0-4 and it is stated that it is a reliable and valid measurement tool for the assessment of fear.
child's anxiety | up to 60 min (when the child wakes up from anaesthetic)
  Child anxiety will be assessed by the "State Anxiety Scale". This scale includes 5 different facial expressions. The children are expected to evaluate how they feel at the moment. Expressions such as "I feel very angry", "I feel angry or" I do not feel angry "are asked to mark the most appropriate one for them.
  The total number of items is 20. The lowest score is 20, the highest the score is 60.
child's pain | up to 60 min (when the child wakes up from anaesthetic)
  Child pain will be assessed by the " Numeric Pain Scale". This method is intended to determine the severity of pain and to explain the patient's pain in numbers. On numerical scales, it starts with the absence of pain (0) and reaches the level of unbearable pain (10).

CONTACTS AND LOCATIONS:
Overall Officials: Timur MEŞE, prof., Study Director — Ministry of Health- İzmir Turkey
Locations (1):
- Dr. Behcet Uz Children's Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Derived] Karakul A, Akgul EA, Yaliniz R, Mese T. Effectiveness of music during cardiac catheterization on children's pain, fear, anxiety and vital signs: A randomized, blind controlled trial. J Pediatr Nurs. 2022 Jul-Aug;65:e56-e62. doi: 10.1016/j.pedn.2022.02.009. Epub 2022 Mar 10. PMID 35279331